CLINICAL TRIAL: NCT06987292
Title: Efficacy of IL-17 Inhibitors on Subclinical Enthesitis in Patients With Moderate to Severe Psoriasis Based on Power Doppler (PD) Ultrasonography (PDUS): a Single-center, Prospective, Exploratory, Open-label Study
Brief Title: A Prospective Study to Assess the Efficacy of IL-17 Inhibitors on Subclinical Enthesitis in Patients With Moderate to Severe Psoriasis Based on Power Doppler (PD) Ultrasonography (PDUS)
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Wenjun HOU, Dr. Wenjun HOU, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2025-0301-02
Record Dates: First submitted 2025-05-05; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis (PsO); Enthesitis; Psoriasis Arthritis; Secukinumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- moderate to severe psoriasis with subclinical enthesitis based on PDUS
  Interventions: Drug: IL-17i

INTERVENTIONS:
Drug: IL-17i — IL-17 inhibitors

SUMMARY:
It is an observational, single-center, prospective, exploratory, open-label study to assess the efficacy and safety of IL-17 inhibitors on subclinical enthesitis in patients with moderate to severe psoriasis with subclinical enthesitis based on Power Doppler (PD) Ultrasonography (PDUS)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( ≥ 18 years of age) with chronic plaque-type psoriasis
2. Meet one of the following conditions: Psoriasis Area and Severity Index [PASI] score > 6, or scalp involvement, or nail involvement.
3. Inflammatory changes on ultrasound consistent with OMERACT definition at least at one peripheral attachment point at screening, defined as thickening and/or abnormal echogenicity of tendons or ligaments at the site of their insertion into the bone (within 2 mm of the talar cortex), and active Doppler signals that may indicate structural damage such as bone erosion, syndesmophytes/calcifications
4. Psoriasis is inadequately controlled by current topical therapy or phototherapy
5. Able to sign the informed consent

Exclusion Criteria:

1. Diagnosis of PsA2 according to CASPAR
2. Any known rheumatic disease, positive rheumatoid factor/anti-citrullinated protein antibodies, prior treatment with anti-rheumatic drugs
3. Treatment with systemic corticosteroids within 12 weeks or 5 half-lives of screening
4. Obesity impeded ultrasound examination
5. Pregnant or lactating women or women with plan for conception 5 months before or after treatment
6. Participated in other clinical trials
7. Concurrent significant medical problems, including but not limited to the following: uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 95 mmHg), congestive heart failure (NYHA class III or IV), total white blood cell count < 2500/μl, or platelets < 100,000/μl or neutrophils < 1500/μl or hemoglobin < 8.5 g/dL at screening.
8. Any liver function abnormality: aspartate aminotransferase (AST) > 2xULN, alanine aminotransferase (ALT) > 2xULN, total bilirubin (TBIL) > 2xULN
9. Abnormal renal function: serum creatinine > 2.0 mg/dl
10. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection, defined as a positive PPD skin test or Mycobacterium tuberculosis interferon-gamma release assay (IGRA) test.
11. Current or relevant history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.
12. History of lymphoproliferative disease, or any known malignancy, or history of malignancy of any organ system within the past 5 years
13. Unable or unwilling to undergo repeated venipuncture
14. History of alcohol or drug abuse or evidence of abuse within 6 months prior to baseline
15. History of hypersensitivity to any component of the study drug
16. Did not accept live vaccines within 4 weeks prior to enrollment, do not have plan of vaccination program during the study, and no live vaccines are planned > 6 months after the last dose of the study (herpes zoster vaccine > 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Glasgow Ultrasound Enthesitis Scoring System (GUESS) from baseline to week 24 | Week 24
  Glasgow Ultrasound Enthesitis Scoring System (GUESS) is an ultrasonographic score of lower limb enthesitis including superior pole of the patella-quadriceps tendon enthesis, inferior pole of the patella-proximal patellar ligament enthesis, tibial tuberosity-distal patellar ligament enthesis, superior pole of the calcaneus-achilles tendon enthesis and inferior pole of the calcaneus-plantar aponeurosis enthesis, composed of assessments of degenerative changes such as tendon thickness, existence of enthesitis, bursitis, or erosions. It is calculated as follows: one point was scored for each abnormality at each site examined, giving a possible maximum total score for both lower extremities 36. A higher score of GUESS represents more serve inflammation and involvement of enthesis while a lower score represents better outcomes.

SECONDARY OUTCOMES:
Change of Glasgow Ultrasound Enthesitis Scoring System(GUESS) from baseline to week 4, 12, 36, 52 | Week 4, 12, 36, 52
  Glasgow Ultrasound Enthesitis Scoring System (GUESS) is an ultrasonographic score of lower limb enthesitis including superior pole of the patella-quadriceps tendon enthesis, inferior pole of the patella-proximal patellar ligament enthesis, tibial tuberosity-distal patellar ligament enthesis, superior pole of the calcaneus-achilles tendon enthesis and inferior pole of the calcaneus-plantar aponeurosis enthesis, composed of assessments of degenerative changes such as tendon thickness, existence of enthesitis, bursitis, or erosions. It is calculated as follows: one point was scored for each abnormality at each site examined, giving a possible maximum total score for both lower extremities 36. A higher score of GUESS represents more serve inflammation and involvement of enthesis while a lower score represents better outcomes.
Complete resolution of enthesitis from baseline to week 24 | Week 24
  Complete resolution of enthesitis from baseline to week 24 based on enthesis assessed by GUESS. It means the percentage reaching a score of 0 for each enthesis. Higher percentage represents higher improvement.
Complete resolution of enthesitis from baseline to week 52 | Week 52
  Complete resolution of enthesitis from baseline to week 52 based on enthesis assessed by GUESS. It means the percentage reaching a score of 0 for each enthesis. Higher percentage represents higher improvement.
New bone erosion, bursitis, osteophytes at week 24 | Week 24
  New bone erosion, bursitis, osteophytes at week 24 based on enthesis assessed by GUESS. It means the percentage that the score changes from 0 to 1 in the item of 'erosion, bursitis, osteophytes' for each enthesis. Higher percentage represents more worsening of inflammation.
New bone erosion, bursitis, osteophytes at week 52 | Week 52
  New bone erosion, bursitis, osteophytes at week 52 based on enthesis assessed by GUESS. It means the percentage that the score changes from 0 to 1 in the item of 'erosion, bursitis, osteophytes' for each enthesis. Higher percentage represents more worsening of inflammation.
Change of patient pain assessment based on Visual Analog Scale (VAS) at week 4, 12, 24, 36, 52 | Week 4, 12, 24, 36, 52
  Change of patient pain assessment based on Visual Analog Scale (VAS) at week 4, 12, 24, 36, 52. The pain VAS is a continuous scale comprised of a horizontal (HVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors. For pain intensity, the scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). Higher score represents more severe pain.
Change of PASI from baseline to week 24, 52 | Week 24, 52
  The Psoriasis Area and Severity Index Score (PASI) is a physician assessment that combines the assessment of the severity (erythema, induration and desquamation) of and area affected by psoriasis into a single score in the range 0 (no disease) to 72 (maximal disease). The higher the score the more severe the psoriasis.
Change of BSA% from baseline to week 24, 52 | Week 24, 52
  Body Surface Area (BSA) is a measure of how much skin is impacted by psoriasis and can be used to track an individual's psoriasis over time. For context, one handprint is equal to approximately 1 percent BSA. Involvement of <3% BSA is considered mild, 3%-10% BSA is considered moderate and >10% of BSA is considered severe psoriasis.
Change of mNAPSI from baseline to week 24, 52 | Week 24, 52
  The mNAPSI is a tool for physicians to evaluate the severity of nail bed psoriasis and nail matrix psoriasis by area of involvement in the nail unit. Each fingernail is rated for the presence and severity of seven features to give a total fingernail score of 0-13 (0= no involvement, 13 = greatest involvement). The total mNAPSI score is the sum of the 10 fingernail scores (range 0-130; 0= no involvement, 130= greatest involvement). The higher the score the more severe the nail bed psoriasis.
Change of PSSI from baseline to week 24, 52 | Week 24, 52
  The Psoriasis Scalp Severity Index scale (PSSI) rates psoriasis severity on the scalp based on three parameters: erythema (redness), scaling, and thickness. Each parameter is assessed individually, and the scores are combined to provide an overall severity rating. The total PSSI score is a sum of scores for erythema, induration, and desquamation x involved area, ranges 0 (no disease) to 72 (maximal disease). The higher the score the more severe the scalp psoriasis is.
Change of HAQ-DI from baseline to week 24, 52 | Week 24, 52
  The HAQ-DI is scored on a four-level difficulty scale ranging from zero (normal, no difficulty) to three (unable to do, extreme difficulty). There are 20 questions covering eight domains: dressing, rising, eating, talking, hygiene, reach, grip, and usual activities. The highest score for an item within each domain is taken as the score for that domain; the HAQ-DI total score is the average of the eight domain scores and therefore ranges between 0 and 3. Scores of 0-1 represent mild to moderate difficulty; 1-2 represent moderate to severe disability; 2-3 represent severe to very severe disability.
Change of SJC66 and TJC68 from baseline to week 24, 52 | Week 24, 52
  66/68 swollen and tender joint counts (SJC66/TJC68)
Change of SPARCC enthesitis index from baseline to week 24, 52 | Week 24, 52
  Medial epicondyle (left/right (L/R)) Lateral epicondyle (L/R) Supraspinatus insertion into greater tuberosity of humerus (L/R) Greater trochanter (L/R) Quadriceps insertion into superior border of patella (L/R) Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R) Achilles tendon insertion into calcaneum (L/R) Plantar fascia insertion into calcaneum (L/R)
Proportion of patients who progressed to PsA at Week 52 | Week 52
  Proportion of patients who progressed to PsA at Week 52, based on CASPAR

OTHER OUTCOMES:
Risk factors at baseline contributing to PsA development | Week 52
  Risk factors at baseline contributing to PsA development (psoriasis phenotype, severity, comorbidities, genetic predisposition, obesity)
Association of risk factors with the development of PsA | Week 52
  Association of risk factors with the development of PsA at 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schett G, Rahman P, Ritchlin C, McInnes IB, Elewaut D, Scher JU. Psoriatic arthritis from a mechanistic perspective. Nat Rev Rheumatol. 2022 Jun;18(6):311-325. doi: 10.1038/s41584-022-00776-6. Epub 2022 May 5. PMID 35513599
- [Background] Chen R, Zhong X, Huang D, Chen Z, Yu Y, Lu J, Wang Q, Kong L, Yi X, Zhao Y, Ding Y, Guo L, Shi Y. Advantages of ultrasound imaging for the early diagnosis of psoriatic arthritis in patients with moderate to severe psoriasis. Heliyon. 2024 Jul 4;10(13):e34136. doi: 10.1016/j.heliyon.2024.e34136. eCollection 2024 Jul 15. PMID 39055795
- [Background] Weiner SM, Jurenz S, Uhl M, Lange-Nolde A, Warnatz K, Peter HH, Walker UA. Ultrasonography in the assessment of peripheral joint involvement in psoriatic arthritis : a comparison with radiography, MRI and scintigraphy. Clin Rheumatol. 2008 Aug;27(8):983-9. doi: 10.1007/s10067-008-0835-y. Epub 2008 Feb 8. PMID 18259687
- [Background] Balint PV, Kane D, Wilson H, McInnes IB, Sturrock RD. Ultrasonography of entheseal insertions in the lower limb in spondyloarthropathy. Ann Rheum Dis. 2002 Oct;61(10):905-10. doi: 10.1136/ard.61.10.905. PMID 12228161